CLINICAL TRIAL: NCT00454857
Title: A Prospective Observational Descriptive Study and Retrospective Chart Review of Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP)
Brief Title: Retrospective & Prospective Observational Study of Patients With Immune (Idiopathic) Thrombocytopenic Purpura (ITP)
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20050237
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Results first posted 2010-05-12 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-10

CONDITIONS: Idiopathic Thrombocytopenic Purpura; Thrombocytopenia; Thrombocytopenia in Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP); Thrombocytopenic Purpura
Keywords: Thrombocytopenia; Chart Review; Platelet; Retrospective; Prospective; Non-interventional; Health Resource Utilization (HRU); Quality of Life (QOL); Immune Thrombocytopenic Purpura (ITP); Idiopathic Thrombocytopenic Purpura (ITP); Immune (Idiopathic) Thrombocytopenic Purpura (ITP); Observational
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia; Purpura, Thrombocytopenic

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: None Retained — None retained.

GROUPS / COHORTS (1):
- Patients with ITP: Participants with ITP and currently treated for ITP were followed prospectively for a period of 12 months.
  Interventions: Other: Retrospective Chart Review; Other: Patient-reported Outcome Questionnaires; Other: Physician Survey

INTERVENTIONS:
Other: Retrospective Chart Review — Retrospective chart review for up to 36 months of enrollment date.
Other: Patient-reported Outcome Questionnaires — Quality of lige questionnaires as well as treatment satisfaction questionnaires are required monthly. Includes QOL, ITP-PAQ (immune thrombocytopenic purpura - patient assessment questionnaire), EQ-5D, and TSQM (Treatment Satisfaction Questionnaire for Medication).
Other: Physician Survey — Physician characteristics to be collected include demographics, years of practice, medical specialty or primary treating physician, and the referral process.

SUMMARY:
This is a multi-center prospective observational descriptive study complemented by a retrospective chart review. Patients diagnosed with ITP and currently treated for ITP by a hematologist or hematologist-oncologist will be recruited from community-based clinics and academic/referral centers. They will be followed prospectively for a period of 12 months. At inception, participants' charts will also be reviewed from the date of enrollment retrospectively to the date of diagnosis or the previous 36 months, whichever is less.

DETAILED DESCRIPTION:
Time Perspective: 12 months prospective chart review study with a retrospective chart review for a period up to 36 months from the start of the study, since the date of diagnosis for ITP.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of ITP according to the American Society of Hematology guidelines (George et al., 1996).
* Is equal to or greater than 18 years of age.
* Is willing and able to complete a series of questionnaires.
* Before any study-specific procedure, the appropriate written informed consent must be obtained.

Exclusion Criteria:

* Participated in clinical trial(s) during the past 36 months.
* Is considering participation in a clinical trial within the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients s diagnosed with ITP and currently treated for ITP by a hematologist or hematologist-oncologist recruited from community based clinics and adademic/referral centers.
Sampling Method: Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2006-05; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: FDA-approved Drug Labeling — http://www.nplate.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With ITP: Patients diagnosed with Immune (Idiopathic) Thrombocytopenic Purpura (ITP) were followed prospectively for a period of 12 months.
Period: Overall Study
Arm/Group | Patients With ITP
Started | 326
Completed Retrospective Chart Review | 324
Completed ≥1 Observational Study Visit | 319
Completed | 272
Not Completed | 54
Not completed — Withdrawal by Subject | 15
Not completed — Lost to Follow-up | 16
Not completed — Noncompliance | 6
Not completed — Death | 5
Not completed — Other | 11
Not completed — Reason unknown | 1

BASELINE CHARACTERISTICS:
Groups:
- Patients With ITP: Patients diagnosed with ITP were followed prospectively for a period of 12 months.
Arm/Group | Patients With ITP
Number analyzed (Participants) | 326
Age Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195
  Male | 131

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Utilizing Immune (Idiopathic) Thrombocytopenic Purpura (ITP) Therapies for First-line Treatment
Description: The number of participants who received ITP therapies for first-line treatment during either the retrospective or prospective phases of the study.
Time Frame: Includes the retrospective chart review (from the date of enrollment retrospectively to the date of diagnosis or the previous 36 months, whichever was less) and the prospective portion of the study (enrollment through Month 12).
Population: All enrolled participants
Measure: Number; unit: Participants
Arm/Group | Patients With ITP
Number analyzed (Participants) | 326
Participants
  Corticosteroids | 128
  IVIG (Intravenous immunoglobulin) | 37
  Rituximab | 3
  Anti-D immunoglobulin | 11
  Splenectomy | 74
  Other | 36

2. Primary Outcome: The Number of Participants Utilizing ITP Therapies for Second-line Treatment.
Description: The number of participants who received ITP therapies for second-line treatment during either the retrospective or prospective phases of the study.
Time Frame: as for outcome 1
Population: All enrolled participants
Measure: Number; unit: Participants
Arm/Group | Patients With ITP
Number analyzed (Participants) | 326
Participants
  Corticosteroids | 98
  IVIG | 54
  Rituximab | 16
  Anti-D immunoglobulin | 16
  Splenectomy | 0
  Other | 48

3. Primary Outcome: The Number of Participants Utilizing ITP Therapies for Third-line Treatment.
Description: The number of participants who received ITP therapies for third-line treatment during either the retrospective or prospective phases of the study.
Time Frame: as for outcome 1
Population: All enrolled participants
Measure: Number; unit: Participants
Arm/Group | Patients With ITP
Number analyzed (Participants) | 326
Participants
  Corticosteroids | 47
  IVIG | 50
  Rituximab | 15
  Anti-D immunoglobulin | 14
  Splenectomy | 0
  Other | 50

4. Primary Outcome: The Number of Participants Utilizing ITP Therapies for Fourth-line Treatment.
Description: The number of participants who received ITP therapies for fourth-line treatment during either the retrospective or prospective phases of the study.
Time Frame: as for outcome 1
Population: All enrolled participants
Measure: Number; unit: Participants
Arm/Group | Patients With ITP
Number analyzed (Participants) | 326
Participants
  Corticosteroids | 26
  IVIG | 28
  Rituximab | 14
  Anti-D immunoglobulin | 14
  Splenectomy | 0
  Other | 56

5. Primary Outcome: The Number of Participants Utilizing ITP Therapies for Fifth-line Treatment
Description: The number of participants who received ITP therapies for fifth-line treatment during either the retrospective or prospective phases of the study.
Time Frame: as for outcome 1
Population: All enrolled participants
Measure: Number; unit: Participants
Arm/Group | Patients With ITP
Number analyzed (Participants) | 326
Participants
  Corticosteriods | 13
  IVIG | 28
  Rituximab | 10
  Anti-D immunoglobulin | 11
  Splenectomy | 0
  Other | 41

6. Primary Outcome: The Number of Participants Utilizing ITP Therapies for Sixth-line Treatment.
Description: Assessed the number of participants who received ITP therapies for sixth-line treatment during either the retrospective or prospective phases of the study.
Time Frame: as for outcome 1
Population: All enrolled participants
Measure: Number; unit: Participants
Arm/Group | Patients With ITP
Number analyzed (Participants) | 326
Participants
  Corticosteriods | 16
  IVIG | 25
  Rituximab | 7
  Anti-D immunoglobulin | 8
  Splenectomy | 0
  Other | 34

7. Primary Outcome: The Number of Participants Utilizing ITP Therapies for Seventh or Greater-line Treatment.
Description: The number participants who received ITP therapies as seventh or greater-line treatment during either the retrospective or prospective phases of the study.
Time Frame: as for outcome 1
Population: All enrolled participants
Measure: Number; unit: Participants
Arm/Group | Patients With ITP
Number analyzed (Participants) | 326
Participants
  Corticosteroids | 30
  IVIG | 33
  Rituximab | 19
  Anti-D immunoglobulin | 11
  Splenectomy | 0
  Other | 41

8. Primary Outcome: The Number of Participants Utilizing ITP Therapies: Treatments With Unknown Starting Date.
Description: The number of participants who received ITP therapies for treatments with unknown starting date during either the retrospective or prospective phases of the study.
Time Frame: as for outcome 1
Population: All enrolled participants
Measure: Number; unit: Participants
Arm/Group | Patients With ITP
Number analyzed (Participants) | 326
Participants
  Corticosteroids | 25
  IVIG | 4
  Rituximab | 0
  Anti-D immunoglobulin | 0
  Splenectomy | 4
  Other | 17

9. Secondary Outcome: Change From Baseline to Month 12 in Quality of Life Measured by the ITP-Patient Assessment Questionnaire (PAQ)
Description: The Immune Thrombocytopenic Purpura Patient Assessment Questionnaire (ITP-PAQ) was developed to assess disease-specific quality of life (QoL) in adults with ITP. It is a 44-item questionnaire that includes scales for physical health (symptoms, fatigue/sleep, bother, and activity), emotional health (psychological and fear), overall QoL, social activity, women's reproductive health, and work. Scores for each scale range from 0 (worst) to 100 (best).
Time Frame: Baseline to month 12 during prospective data collection phase
Population: The Patient Reported Outcome (PRO) Analysis Set includes all participants who completed at least one questionnaire during the prospective observation period.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patients With ITP
Number analyzed (Participants) | 274
Units on a scale
  Physical Health-Symptoms score | 6.7 (17.1)
  Physical Health - Fatigue score | 7.2 (23.7)
  Physical Health - Bother score | 9.4 (22)
  Physical Health - Activity score | 9 (24.5)
  Emotional Health - Psychological score | 6.4 (21.2)
  Emotional Health - Fear score | 4 (16)
  Quality of Life score | 9.2 (21.9)
  Social Quality of Life score | 3.4 (15.5)
  Woman's Reproductive Health (WRH) score | 4.7 (17)
  WRH: Menstrual Symptoms score | 5.9 (22.4)
  Woman's Reproductive Health: Fertility score | 4.2 (19)
  Work Quality of Life score | 3.8 (14)

10. Secondary Outcome: Change From Baseline to Month 12 in Health-related Quality of Life Assessed by EuroQol Visual Analog Scale (EQ-5D VAS)
Description: The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' (score = 100) and 'Worst imaginable health state' (score = 0).
Time Frame: Baseline to Month 12 during prospective data collection phase
Population: The Patient Reported Outcome (PRO) Analysis Set includes all subjects who completed at least one questionnaire during the prospective observation period.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patients With ITP
Number analyzed (Participants) | 274
Units on a scale | 4.1 (18.00)

11. Secondary Outcome: Change From Baseline to Month 12 in Treatment Satisfaction
Description: Participant satisfaction with treatment was measured using the Treatment Satisfaction Questionnaire for Medication (TSQM), an 11-item questionnaire providing scores on four scales - side effects, effectiveness, convenience and global satisfaction. TSQM Scale scores range from 0 to 100 with higher scores indicating more satisfaction with treatment.
Time Frame: Baseline to Month 12 during prospective data collection phase
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patients With ITP
Number analyzed (Participants) | 274
Units on a scale
  Overall Satisfaction score | 1.8 (19.40)
  Efficacy score | 2.8 (21.02)
  Side Effects score | 7.9 (20.79)
  Convenience score | 0.3 (17.74)

12. Secondary Outcome: Number of Participants Receiving Drug Therapies for Treatment of ITP During the Prospective Phase
Description: The number of participants who received drug therapies for the treatment of ITP during the prospective phase of the study. Use of multiple medications by the same participants is possible.
Time Frame: 12 months (prospective data collection phase)
Population: All enrolled participants who completed at least 1 observational study visit during the prospective phase.
Measure: Number; unit: Participants
Arm/Group | Patients With ITP
Number analyzed (Participants) | 319
Participants
  Anti-D | 14
  Azathioprine | 14
  Corticosteroids-IV (Intravenous) | 7
  Corticosteroids-Oral | 49
  Cyclophosphamide | 4
  Danazol | 19
  IVIG | 42
  Rituximab | 25
  Vincristine/Vinblastine | 1
  Other | 43

13. Secondary Outcome: Duration of Exposure to ITP Medication
Description: Duration of exposure to each ITP medication measured from enrollment until the end of the 12-month data collection phase.
Time Frame: 12 months (prospective data collection phase)
Population: All enrolled participants who completed at least 1 observational study visit during the prospective phase. N=number of participants using each medication.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Patients With ITP
Number analyzed (Participants) | 319
Months
  Anti-D immunoglobulin (N=14) | 2.0 (3.90)
  Azathioprine (N=13) | 7.3 (5.18)
  Corticosteriods-Intravenous (N=7) | 0.2 (0.41)
  Corticosteriods-Oral (N=37) | 3.6 (3.78)
  Cyclophosphamide (N=4) | 1.5 (1.59)
  Danazol (N=18) | 7.5 (4.27)
  Intravenous immunoglobulin (N=41) | 0.7 (2.00)
  Rituximab (N=24) | 0.7 (0.44)
  Vincristine/Vinblastine (N=1) | 0.0 (NA) — Only 1 participant with data
  Other (N=42) | 6.6 (6.57)

14. Secondary Outcome: Number of Participants Requiring Splenectomy
Description: The number of participants who required a splenectomy during the 12-month prospective phase of the study.
Time Frame: 12 months
Population: All enrolled participants who completed at least 1 observational study visit during the prospective phase.
Measure: Number; unit: Participants
Arm/Group | Patients With ITP
Number analyzed (Participants) | 319
Participants | 15

ADVERSE EVENTS:
Description: No AEs were collected for this protocol
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.